CLINICAL TRIAL: NCT07243639
Title: A Prospective Study on the Efficacy and Safety of a Novel Oral Drug, Etrasimod, in Elderly Patients With Ulcerative Colitis
Brief Title: Efficacy and Safety of Etrasimod in Elderly Patients With Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Etrasimod in elderly UC
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis (Disorder)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elderly patients (aged 65 years or older) with active ulcerative colitis (Experimental)
  Interventions: Drug: Etrasimod administration

INTERVENTIONS:
Drug: Etrasimod administration — 2 mg of Etrasimod is orally administered everyday.

SUMMARY:
Eligible patients will be identified in regular clinical practice. After providing thorough explanation and obtaining voluntary written informed consent, the clinical course, adverse events, endoscopic findings, and histopathological changes in biopsy specimens after Etrasimod administration will be prospectively collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active ulcerative colitis

Exclusion Criteria:

* the presence of acute or chronic renal failure, chronic heart disease, pulmonary infection, liver cirrhosis, colorectal cancer, autoimmune disease, and infectious disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: Clinical remission rate at 4 weeks (Clinical activity Index score <4) (max.29, min. 0) | 4 weeks

SECONDARY OUTCOMES:
Secondary endpoints: Endoscopic improvement rate at 52 weeks (Mayo Endoscopic Subscore (MES) <1 or improved (Ulcerative colitis endoscopic of severity, UCEIS), and incidence of adverse events during the study | 52 weeks
  MES: Min. 0, Max 3, UCEIS: Min. 0, Max 8

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: Undecided